CLINICAL TRIAL: NCT00501020
Title: A 24-Week Randomized, Double-blind, Double-Dummy, Multicenter Study to Compare the Efficacy of AVANDIA When Added to Submaximal Doses of Metformin and to Compare the Tolerability of the Combination to Metformin Monotherapy When Administered to Subjects With Type 2 Diabetes Mellitus
Brief Title: Comparison of the Efficacy and Tolerability of the Addition of AVANDIA to Submaximal Doses of Metformin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 49653/284
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; metformin; rosiglitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rosiglitazone

SUMMARY:
This was a randomized, double-blind, double dummy, multicenter study to assess the safety, efficacy and tolerability of the addition of RSG (rosiglitazone) to sub-maximal MET (metformin) combination relative to maximal MET monotherapy in subjects with type 2 DM (diabetes mellitus). The total duration of the study was approximately 20 months. The study consisted of a two-week washout period, a four to seven-week MET titration period, and a 24-week randomized treatment phase in which subjects, stratified by prior therapy, received either RSG + MET combination therapy or MET monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of Type 2 DM as defined by the criteria of the American Diabetes Association.
* Exceptions were granted to those subjects over the age of 75 on a case-by-case basis and only with the expressed permission of the study sponsor.
* Females who were post-menopausal (i.e., >6 months without a menstrual period), surgically sterile, or using acceptable contraceptive measures (oral contraceptive, Norplant, Depo-Provera, an IUD, a diaphragm with spermicide or condoms).
* Subjects previously treated by either diet and exercise or oral therapy. Any subjects who were receiving MET or MET plus Sulfonylurea (SU) must have been receiving no more than MET 1000mg/day for at least three months prior to study entry. Subjects must have stopped previous treatment with thiazolidinediones (TZDs) at least three months prior to screening.
* Subjects with a Body Mass Index (BMI) >=27 kg/m2.
* Subjects who signed the Informed Consent.
* Subjects who received monotherapy treatment within the last three months prior to study entry or drug-naives who had HbA1c levels between 7% and 10%, inclusive. Subjects who received prior combination treatment had HbA1c of at least 6.5% to 8.5%, inclusive.
* Subjects with FPG of <270 mg/dL at screening and visit 2, must have had a FPG >=126 mg/dL at either screening or at the MET titration period (visit 2, run-in) for entry into the treatment phase of the study.

Exclusion Criteria:

* Females who were lactating, pregnant, or planning to become pregnant.
* Any clinically significant abnormality identified on the chest X-ray, screening physical examination, laboratory tests, or electrocardiogram, which, in the judgment of the investigator, would preclude safe completion of the study.
* Use of TZDs or any investigational drug for glycemic control within three months prior to study entry irregardless of the treatment regimen, or use of any other investigational agent (not related to glycemic management) within 30 days or five half-lives (whichever is longer) preceding study entry.
* Subjects with FPG >=270 mg/dL at screening.
* Subjects with prior history of hepatocellular reaction to or severe edema associated with troglitazone or any current TZD.
* History of significant hypersensitivity to TZDs, biguanides, or compounds with similar chemical structures.
* Subjects currently using insulin or who discontinued its use for glycemic control within the last three months prior to study entry.
* History of acute or chronic metabolic acidosis.
* Presence of clinically significant renal or hepatic disease (i.e., male subjects with serum creatinine >1.5 mg/dL; female subjects with serum creatinine >1.4 mg/dL; ALT, AST, total bilirubin, GGT, or alkaline phosphatase >2.5 times the upper limit of the reference range).
* Anemia defined by hemoglobin concentration <11.0 g/dL for males or <10.0 g/dL for females.
* Presence of unstable or severe angina or coronary insufficiency, or any congestive heart failure requiring pharmacologic treatment.
* Systolic BP >170mmHg or diastolic BP >100mmHg while on anti-hypertensive treatment.
* Recent history or suspicion of current drug abuse or alcohol abuse (defined as the consumption of more than 35 units of alcohol per week.
* Non-compliance with study medication during MET titration period (run-in).
* Subjects, who received or anticipated receiving radiocontrast dye during the MET titration (run-in) or the randomized treatment period of the study.
* Subjects unwilling or unable to comply with the procedure described in the protocol.
* Subjects who were unable to read or understand the English language were excluded from the study due to the administration of the QOL assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750
Dates: Start 2001-06-05 (Actual); Primary Completion 2003-02-13 (Actual); Study Completion 2003-02-13 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable was HbA1c change from baseline (visit 3) after 24 weeks of treatment with either RSG+MET combination therapy or Metformin monotherapy. | 24 Weeks

SECONDARY OUTCOMES:
Secondary efficacy variables included: the change from baseline (visit 3) at week 24 (visit) in FPG, immunoreactive insulin, HbA1c and FPG responders, Questionnaire-Tolerability of GI side-effects, and Questionnaire - Quality of Life. | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Goldstein BJ, Cobitz AR, Hand LM, Chen H. Are the metabolic effects of rosiglitazone influenced by baseline glycaemic control? Curr Med Res Opin. 2003;19(3):192-9. doi: 10.1185/030079903125001695. PMID 12803733
- [Result] Rosenstock J, Goldstein BJ, Wooddell MJ, Strow LJ, Waterhouse BR, Cobitz AR Greater benefits of rosiglitazone added to submaximal dose of metformin compared to maximizing metformin dose in type 2 diabetes mellitus patients. Diabetes 2004; 53 (Suppl 2): A144 Poster presented at ADA
- [Result] Weissman PW, Goldstein BJ, Campbell JC, Gould ER, Waterhouse BR, Strow LJ, Cobitz AR. Rosiglitazone plus metformin combination effects on CV risk markers suggest potential CV benefits in type 2 diabetes patients. Diabetes 2004;53(Suppl 2): A28 Oral presentation at ADA
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 49653/284 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 49653/284 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 49653/284 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 49653/284 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 49653/284 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 49653/284 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 49653/284 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register